CLINICAL TRIAL: NCT03985228
Title: Promotion of Consumer's Health: Nutritional Enhancement/Valorization of Agrofood Italian Traditional Products (PROS.IT)
Brief Title: Nutritional Trial With Probiotic Fortified Milk in Women Affected by Insomnia
Acronym: Prosit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Claudio Franceschi, Professor emeritus, University of Bologna
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MIUR prot.n.257/Ric.
Record Dates: First submitted 2016-07-22; First posted 2019-06-13 (Actual); Last update posted 2019-06-13 (Actual); Status verified 2019-06

CONDITIONS: Sleep Disorders
Keywords: golden milk, insomnia, gut-brain axis
MeSH Terms: conditions — Sleep Wake Disorders; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fortified milk (Experimental): The subjects assumed daily 250 ml of fortified milk for 12 weeks.
  Interventions: Dietary Supplement: Fortified milk
- Placebo milk (Placebo Comparator): The subjects assumed daily 250 ml of placebo milk for 12 weeks.
  Interventions: Dietary Supplement: Placebo milk

INTERVENTIONS:
Dietary Supplement: Fortified milk — Ultra high temperature UHT, partly-skimmed milk (1% fat), highly digestible (lactose <0.01%), enriched in whey protein (5%) and calcium (0.24%), supplemented with unsaturated fatty acids omega-3 (DHA + EPA), vitamins (D, B12, B6, B9, E, C), prebiotics (FOS) and phyto curcuminoids (sunflower lecithin). Milk had to be associated with a packet of lyophilized and concentrated probiotics (Bifidobacteria infant-type and / or Lactobacilli), at the time of consumption. Milk and probiotics had been produced or supplied by Granarolo s.p.a.
  Other Names: golden milk
  Arms: Fortified milk
Dietary Supplement: Placebo milk — Ultra high temperature UHT, partly-skimmed milk (1% fat), highly digestible (lactose <0.01%) with standard proteins of milk (3.1%) and color additive "quantum satis". Milk had to be associated with a packet of maltodextrin "Food Grade", at the time of consumption. Milk and maltodextrin had been produced or supplied by Granarolo s.p.a.
  Arms: Placebo milk

SUMMARY:
The study "Nutritional Trial With Probiotic Fortified Milk in Women Affected by Insomnia" is a part of a complex and multi-sectoral development research project (PROS.IT) with the participation of University Research Institutes and small/medium Italian enterprises.

The general objective of the Project is to promote the collaboration between the best scientific research, both epidemiological and experimental, and the most advanced technologies to develop fortified foods that meeting the specific nutritional requirements of adult consumers. This objective will be achieved by the nutritional improvement of primary production, the development of innovative functional foods at high added value, in addition to traditional products functionalized, which are peculiar of the Italian local districts.

DETAILED DESCRIPTION:
Sleep disorders and, in particular, insomnia, are quite common conditions in over 55 population, especially among women. Insomnia becomes a chronic pathology when the difficulty in initiating or maintaining sleep occurs more times a week for several months and is associated to a constant feeling of fatigue, concentration problems, mood disorders and social and family troubles severely impairing the quality of life. In according to the sleep hygiene guidelines, the therapeutic treatments for insomnia include drugs (benzodiazepines, non-benzodiazepines, antidepressants) with often not fully satisfactory results for the patient and entailing a series of side effects, such as daytime sleepiness, lack of attention and energy in addition to mental confusion. Recently, some researches in neurological field have shown that disorders affecting central nervous system, as well as sleep and circadian rhythm disruption, can be associated to specific alteration of the gut microbiota. The enteric nervous system has been referred to as a "second brain" able to interact with the central nervous system impinging upon higher cognitive functions through a bidirectional communication system known as gut-brain axis. The gut microflora plays a crucial role in gut-brain axis, modulating stress response through the Hypothalamic-Pituitary-Adrenal axis and thus influencing memory, mood, cognition and sleep architecture. Therefore, a non-pharmacological intervention aimed to improve gut microbiota and the inflammatory bowel conditions could be an effective strategy to counteract insomnia. In the framework of Pros.IT project, the Granarolo S.p.A. in collaboration with the University of Bologna has developed a milk enriched with different micronutrients (vitamins, ω-3 fatty acids, prebiotics, curcumin) and "infant-type" probiotics isolated from human milk and endowed with immunomodulating activity. This supplementation should improve the overall health status, and in particular the plant extracts, prebiotics and probiotics with anti-inflammatory and immunomodulatory activities should ameliorate significantly sleep quality and stress perception through the modulation of gut microbiota and gut-brain axis.

The main goal of this study is to evaluate the effect of the administration of a functional milk reinforced with probiotics (250ml/die), vitamins and other micronutrients on sleep of patients suffering from chronic insomnia. An objective assessment it requires a value at least higher than 3% of increase of the sleep efficiency, since the 3% is the percentage of improvement recognized to the common drugs against insomnia. The study is randomized, double-blind, placebo-controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with an age between 55 and 70 years old, only females, free-living, affected by chronic insomnia defined according to the criteria of the International Classification of Sleep Disorders (2014).

Exclusion Criteria:

* Allergy or intolerance to cow's milk. Use of Benzodiazepines, "Z drugs" or anti-depressive drugs during the three months preceding the start of the trial. Celiac disease and other intestinal malabsorption or inflammatory bowel diseases (Crohn's disease and ulcerative colitis). Chronic therapy with anticoagulant, corticosteroid, anticancer drugs and immunosuppressants. Diabetes type I and type II, chronic viral hepatitis, neurological disorders or dementia, cancer, poor prognosis disease in the short term. Use of anti-inflammatory drugs or inflammatory-infective events within 7 days before the start of the trial and use of antibiotics or vaccinations within 30 days before.

Ages: 55 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-11-20; Primary Completion 2016-07 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Self reported quality of sleep | Change from baseline Sleep evaluation at 12 weeks milk intake
  Sleep quality assessed by questionnaires
Measured quality of sleep | Change from baseline Sleep evaluation at 12 weeks milk intake
  assessed by actigraph

SECONDARY OUTCOMES:
Levels of stress | 12 weeks
  Stress was evaluated by PSS questionnaire and 24-h urinary cortisol levels
Inflammatory status | 12 weeks
  Dosage in plasma of the following cytokines: IL-1β, IL-4, IL-6, IL-10, IL-17A, IL-17F, IL-21, IL-22, IL-23, IL-25, IL-31, IL-33, IFN-γ, sCD40L, TNF-α, IL-17 A/F by Elisa immunoassay.
Evalution of glycomics | 12 weeks
  Plasmatic N-glycans by capillary electrophoresis (DSA-FACE).
Levels of anxiety | 12 weeks
  Stress was evaluated by STAI-Y2
Levels of depression. | 12 weeks
  Stress was evaluated by BDI-II questionnaire
Evalution of epigenetic | 12 weeks
  Epigenetic analysis of ELOVL2, FHL2, PENK genes by "Sequenom"
Gut Microbiota composition | 12 weeks
  Analysis of gut-microbiota composition by 454 Pyrosequencing of the V4 region of the 16S rRNA gene.

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Franceschi, MD, Principal Investigator — University of Bologna
Locations (1):
- University of Bologna-Department of Speciality, Diagnostic and Experimental Medicine, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No